CLINICAL TRIAL: NCT00750984
Title: A Comparison of Two Different Surgical Techniques for Total Hip Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU9
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2016-09

CONDITIONS: Arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This arm utilizes the anterolateral approach using the ReCap® Total Hip Resurfacing System.
  Interventions: Procedure: Anterolateral approach; Device: ReCap Total Hip Resurfacing
- 2 (Active Comparator): This arm utilizes the posterior approach using the ReCap® Total Hip Resurfacing System.
  Interventions: Procedure: Posterior approach; Device: ReCap Total Hip Resurfacing

INTERVENTIONS:
Procedure: Anterolateral approach — The anterolateral approach is performed with the patient positioned on the side. The blood supply to the femoral neck from the medial circumflex artery is regarded preserved by this surgical method.
  Arms: 1
Procedure: Posterior approach — The posterior approach is performed with the patient positioned on the side. The medial circumflex artery is cut at the lower border of the short external rotators risking a compromised blood supply to the femoral head.
  Arms: 2
Device: ReCap Total Hip Resurfacing — This arm utilizes the anterolateral approach using the ReCap® Total Hip Resurfacing System.
  Arms: 1
Device: ReCap Total Hip Resurfacing — This arm utilizes the posterior approach using the ReCap® Total Hip Resurfacing System.
  Arms: 2

SUMMARY:
This study compares the posterior approach to the anterolateral approach using the ReCap® Total Hip Resurfacing System.

DETAILED DESCRIPTION:
Theoretical considerations of RECAP procedures through anterolateral trochanteric osteotomy:

* Less bone resection, less complicated revision surgery.
* Reduced stress shielding of the femur.
* Lower incidence of hip dislocations.
* Walking function improved by change in mobilisation regime and operative technique.
* Risk of femoral neck fracture is reduced by preoperative measurement of bone density.
* Risk of avascular necrosis of the femoral head is reduced with the anterolateral approach preserving femoral head blood supply and preventing later failure of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip OA
* Secondary hip OA due to mild and moderate acetabular dysplasia
* Sufficient bone quality for cementless acetabular component
* Suited for resurfacing of the femoral head (pre- and intraoperatively assessed)
* >29 years
* <61 years

Exclusion Criteria:

* Neuromuscular or vascular diseases in affected leg
* Patients found intra-operatively to be unsuited for a cementless acetabular component or cementing of the femoral component
* Need of NSAID post-operatively
* Fracture sequelae
* Females at risk of pregnancy (no safe contraceptives)
* Severe hip dysplasia
* Sequelae from hip disease in childhood
* Medicine with large effect on bone density (K-vitamin antagonists, loop-diuretic)
* Alcoholism (females > 14 units per week, males > 21 units per week) AVN
* Osteoporosis

Ages: 29 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
RSA | 1 week, 3 months, 1 year, 2 years, 5 years

SECONDARY OUTCOMES:
Harris Hip Score | Pre-operatively, 1 week, 6 weeks, 3 months, 1 year
Microdialysis | 1 week
Conventional X-ray | 1 week
Gait Analysis | 1 week, 3 months, 1 year
DEXA scan | Pre-operatively, 1 week, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pryno, MD, Principal Investigator — Aarhus University Hospital; Kjeld Soeballe, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark